CLINICAL TRIAL: NCT01004952
Title: Measuring Real Time Decision-Making About UVR Protection
Brief Title: Measuring Real Time Decision-Making About Ultraviolet Radiation (UVR) Protection
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of British Columbia (Other); San Diego State University (Other); Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-137
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Skin; Sunscreen; UVR Protection; 09-137
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- screening questionnaire: This study will involve two phases. Guided by EDTM, we will first build models of decision-making about UVR protection (sunscreen use, shade-seeking, hat use, use of protective clothing)using in-home ethnographic interviews with 25 melanoma FDRs (Phase I). In Phase II, we will test the validity of each composite model. This will be completed using EMA data collection with 60 different melanoma FDRs from Phase I who will report on their sunscreen use, shade-seeking, use of hat, and use of UVR protective clothing and decision-making regarding these outcomes via interactive voice response (IVR) system and audio narrative diaries (using a digital voice recorder). We will examine the validity of each model and examine the influence of theory-driven affective and cognitive predictors of UVR protection maintenance across time.
  Interventions: Behavioral: screening questionnaire

INTERVENTIONS:
Behavioral: screening questionnaire — Phase I involves in-home interviews of 25 participants to understand the factors that affect participants' decision-making about UVR protection (sunscreen use, shade-seeking, hat use, use of protective clothing). In Phase II, we plan to recruit a sample of 60 melanoma first degree relatives (FDRs) and use an electronic narrative diary to record their daily behaviors about UVR protection. They will be asked to carry a interactive voice response (IVR) system for 14 days and they should be in the continental United States.

SUMMARY:
The purpose of this study is to understand how people make decisions about sun protection. This study is important in helping to protect against sun exposure, since it is a main risk factor for melanoma. The investigators would like to understand the decisions people make about sun protection so that they can improve their ability to help individuals who may be at risk for melanoma.

ELIGIBILITY:
Inclusion Criteria:

* A first-degree biological relative (a child, sibling or parent) as per self report of an MSKCC follow-up surgical patient diagnosed with melanoma as per pathology report or clinician's judgment;
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.
* 18 years of age or older;
* For Phase I only: FDRs who live within a 50 mile radius of MSKCC to make it feasible for Ms. Shuk to be able to arrive at each person's home for the in-home interview without the cost being prohibitive;
* For Phase I only: Can recall a period when s/he was out in the sun for at least one hour on a sunny day this past summer 2009.
* For Phase I only: Can recall a separate period when s/he was out in the sun for at least one hour on a sunny day this past summer 2009, but s/he was in a different location from the period referenced above.
* For Phase II only: FDRs who self-report at least 1 consecutive hour in the morning (dawn to 12:30pm) and 1 consecutive hour in the afternoon (12:30-5pm) of daily (weekend and weekday) outdoor activities on the screening questionnaire

Exclusion Criteria:

* First-degree relatives of melanoma patients who report never using UVR protection;
* Patient's who provide consent for Phase I will not be eligible for Phase II.
* Any first-degree relative of a melanoma patient who already has a first-degree relative who consented to the study;
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients whose FDRs may be eligible for this study will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC) will identify patients who are melanoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2009-10-27 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hay, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Phase I: 25 Melanoma FDRs; Phase II: 60 Melanoma FDRs: This study will involve two phases. Guided by EDTM, we will first build models of decision-making about UVR protection (sunscreen use, shade-seeking, hat use, use of protective clothing)using in-home ethnographic interviews with 25 melanoma FDRs (Phase I). In Phase II, we will test the validity of each composite model. This will be completed using EMA data collection with 60 different melanoma FDRs from Phase I who will report on their sunscreen use, shade-seeking, use of hat, and use of UVR protective clothing and decision-making regarding these outcomes via interactive voice response (IVR) system and audio narrative diaries (using a digital voice recorder). We will examine the validity of each model and examine the influence of theory-driven affective and cognitive predictors of UVR protection maintenance across time.
  screening questionnaire: Phase I involves in-home interviews of 25 participants to understand the factors that affect participants' decision-making about UVR protection (sunscreen use, shade-seeking, hat use, use of protective clothing). In Phase II, we plan to recruit a sample of 60 melanoma first degree relatives (FDRs) and use an electronic narrative diary to record their daily behaviors about UVR protection. They will be asked to carry a interactive voice response (IVR) system for 14 days and they should be in the continental United States.
Period: Overall Study
Arm/Group | Cohort 1: Phase I: 25 Melanoma FDRs | Phase II: 60 Melanoma FDRs
Started | 25 | 69
Completed | 25 | 53
Not Completed | 0 | 16
Not completed — Lost to Follow-up | 0 | 11
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Phase I: 25 Melanoma FDRs | Phase II: 60 Melanoma FDRs | Total
Number analyzed (Participants) | 25 | 59 | 84
Age, Continuous [Mean (Full Range); unit: years] | 39 [19 to 78] | 48 [18 to 82] | 45 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 38 | 50
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 57 | 81
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 58 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 59 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Interviewed on UVR Protection Behaviors.
Description: To generate models explaining decision-making about four UVR protection behaviors (sunscreen use, shade-seeking, hat use, use of protective clothing) in melanoma FDRs. This was an inductive, qualitative study using an open-ended interview to accomplish the Aim. Cohort 1 was used for this Aim.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Phase I: 25 Melanoma FDRs | Phase II: 60 Melanoma FDRs
Number analyzed (Participants) | 25 | 59
Participants
  Number of participants interviewed | 25 | 0
  Number of participants not interviewed | 0 | 59

2. Secondary Outcome: To Examine Theory-driven Affective and Cognitive Predictors of UVR Protection Maintenance (Sunscreen Use, Shade-seeking, Hat Use, and Use of UVR Protective Clothing)Assessed in Real Time.
Description: To examine theory-driven affective and cognitive predictors of UVR protection maintenance (sunscreen use, shade-seeking, hat use, and use of UVR protective clothing) assessed in real time. Phase 1 was not assessed for this Outcome Measure.
Time Frame: 1 year
Population: Phase 1 was not assessed for this Outcome Measure
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Phase I: 25 Melanoma FDRs | Phase II: 60 Melanoma FDRs
Number analyzed (Participants) | 0 | 59
Participants
  Women who use sunscreen in cooler weather: number analyzed (Participants) | 0 | 38
  Women who use sunscreen in cooler weather | 0 | 9
  Men who skip sunscreen in cooler weather and in shade while wearing a hat: number analyzed (Participants) | 0 | 21
  Men who skip sunscreen in cooler weather and in shade while wearing a hat | 0 | 21
  Women who skip sunscreen in cooler weather and in shade while wearing a hat: number analyzed (Participants) | 0 | 38
  Women who skip sunscreen in cooler weather and in shade while wearing a hat | 0 | 23
  Men who skip sunscreen on sunny days and in shade while wearing a hat: number analyzed (Participants) | 0 | 21
  Men who skip sunscreen on sunny days and in shade while wearing a hat | 0 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1: Phase I: 25 Melanoma FDRs | Phase II: 60 Melanoma FDRs
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/59
Other Adverse Events (participants affected / at risk) | 0/25 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT01004952/Prot_SAP_000.pdf